CLINICAL TRIAL: NCT01418079
Title: Accuracy of the O2 MedTech PMS-3000 Monitor for the Non-invasive Measurement of Cerebral and Tissue Oxygenation Using Phase-modulated Infrared Spectroscopy
Brief Title: Accuracy of the O2 MedTech PMS-3000 Monitor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: O2 MedTech, Inc. (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2010001
Record Dates: First submitted 2011-08-12; First posted 2011-08-16 (Estimated); Last update posted 2012-05-23 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Spectroscopy, near infrared; cerebral oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PMS-3000 (Experimental): Human volunteers undergo oxygen desaturation in order to determine the accuracy of the device over a clinical range of oxygen saturations 70 - 100%.
  Interventions: Device: O2 MedTech cerebral oximeter (Oxygen desaturation)

INTERVENTIONS:
Device: O2 MedTech cerebral oximeter (Oxygen desaturation) — Reduction in blood oxygen saturation by sequential reduction in inspired gas composition. Steps are of 6 minutes duration with reduction in pulse oximeter oxygen saturation from 100 to 70%.
  Other Names: PMS-3000 cerebral oximeter

SUMMARY:
A cerebral oximeter is a device that uses light to measure the amount of oxygen within the brain. It is similar to the device that measures the level of oxygen in the tip of the finger, known as a pulse oximeter. The cerebral oximeter consists of a sensor placed on the forehead that both emits and detects the amount of light absorbed. This study will determine how accurate the device is by comparing the displayed value on the monitor with blood samples taken simultaneously from the arterial blood in the wrist and venous blood in the neck. In order to test the device over a suitable range, the level of oxygen within the blood will be reduced in a controlled manner by reduction of the inspired oxygen concentration. This is the equivalent of ascending to an altitude of 16,000 feet. The study will be conducted in healthy volunteers.

DETAILED DESCRIPTION:
This is a calibration and validation study of a near-infrared spectroscopy (NIRS) device designed to measure the cerebral tissue oxygen saturation non-invasively. This is achieved by comparing NIRS-derived cerebral tissue oxygen saturation with a calculated value derived from simultaneous arterial and jugular venous blood samples.

At present the FDA have adopted the standards published in 2005 by the International Organization for Standardization (ISO), entitled ISO 9919. This is a set of technical specifications and guidelines for pulse oximeters, which share certain technical similarities to cerebral oximeters. In particular, Annex EE details the conduct of a controlled desaturation study for the calibration of pulse oximeter equipment. Specifically, the fraction of inspired oxygen delivered to test subjects is varied to achieve a series of targeted steady state saturation periods over a range of arterial oxygen saturation of 70 - 100%.

While cerebral oximeters differ from pulse oximeters in terms of the what is being measured (brain tissue versus arterial blood) the FDA have maintained the requirement to examine data from human volunteer studies in which the arterial oxygen saturation ranges from 70 - 100%. Several FDA-approved cerebral oximeters were validated in a similar manner.

The device controlling the inspired gas concentration is the RespirAct, which permits precise reduction in the arterial oxygen saturation while also maintaining the arterial carbon dioxide level at a precise level.

The study consists of 2 sequences:

* First sequence: reduction in arterial oxygen saturation in approximately 5% increments from 100 to 70%, while maintaining the arterial carbon dioxide level at 40 mmHg, followed by return to room air and then a period of supplemental oxygen.
* Second sequence: reduction in arterial oxygen saturation in approximately 5% increments from 100 to 70%, while maintaining the arterial carbon dioxide level at a different level, followed by return to room air and then a period of supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

1. Body Mass Index (BMI) of 18 to 30, inclusive
2. No anticoagulant or platelet inhibitor use
3. Oxygen saturation (SpO2) ≥ 95% on room air
4. Able to tolerate breathing mask apparatus

Exclusion Criteria:

1. Female with positive pregnancy test
2. Beard or history of or anatomy suggestive of difficult airway
3. Lab values outside normal range for the clinical site
4. History of cigarette smoking or currently a cigarette smoker
5. Current drug or alcohol abuse
6. History of sleep apnea, high blood pressure (HBP), cardiac or pulmonary disease, gastroesophageal reflux, hemoglobinopathy, or coagulation abnormality
7. Known allergy to lidocaine or heparin
8. Abnormal electrocardiogram (ECG)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2011-08; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Accuracy of device to measure cerebral tissue oxygen saturation | approximately 4 months
  Oximeter measurements are compared to co-oximeter measurements following each subject study. The total sample of subjects is needed to complete the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: David B MacLeod, FRCA, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States